CLINICAL TRIAL: NCT03927755
Title: REASON 2 Trial - Timing For Single View Bedside Cardiac Ultrasound
Brief Title: Timing For Single View Bedside Cardiac Ultrasound
Acronym: REASON-2
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Romolo Gaspari, Professor, Department of Emergency Medicine, University of Massachusetts, Worcester
Other Study IDs: UMASS-ED-4-22-19
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Echocardiography
Keywords: Bedside Ultrasound
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sub-xyphoid: Ultrasound views of the heart obtained using the sub-typhoid approach. Individuals with a mix of co-morbidities but are clinically stable will be viewed. Physicians with experience in bedside ultrasound are being studied.
  Interventions: Other: Education
- Para-sternal Long: Ultrasound views of the heart obtained using the parasternal long approach. Individuals with a mix of co-morbidities but are clinically stable will be viewed. Physicians with experience in bedside ultrasound are being studied.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Physicians will undergo training on how to rapidly obtain appropriate images.

SUMMARY:
The goal of this study is to measure the hypothetical minimal amount of time it takes to perform a single view bedside trans-thoracic echo (TTE) comparing sub-xyphoid view and the parasternal long view. Physicians will be timed from initiation of imaging to completion of the recording of a single view of the heart. Images will be rated for quality.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational trial involving sites across the United States and Canada. Residents will be enrolled when performing ultrasound imaging on non-critically ill patients in the emergency department. Residents obtaining cardiac ultrasound images on patients in the emergency department during pre-planned educational sessions will be enrolled in a prospective manner.

Physicians participating in this study will undergo a short educational session on both techniques of cardiac ultrasound as well as rationale for performing cardiac ultrasound rapidly during cardiac arrest. This educational intervention will provide the cognitive framework for the physicians to participate in the study. Physicians will be told to obtain the images as fast as possible and to get good quality images but they will be able to stop imaging if they are unable to obtain the images rapidly.

Individual physicians will be randomized to obtain a single parasternal or sub-xyphoid view of the hear first, followed by the other view. TTE will be performed on conscious and awake patients in the emergency department. Imaging will be performed in front of research staff. Primary outcome is time from transducer-skin contact to completion of the digital recording of a visible heart beating. Secondary outcome is the quality of the ultrasound image using a 5-point image quality scale.

Patients who will be imaged in this study will be those patients that would have been imaged during the existing educational session (scan shift). The patient will not need consent but can be told about the study if needed. No patient will be imaged if they have the possibility of having a clinical deterioration during the ultrasound imaging. Each set of images (PSL and SX) will be from a unique patient.

Subject data, with Protected Health Information (PHI) removed, will be recorded on data sheets prior to uploading into a centralized electronic database as soon as possible. Data will be obtained during the educational encounter including: Resident ID, post graduate year (PGY) level, Number of Cardiac Ultrasounds performed prior to starting study, US view attempted first, Imaging duration (seconds), Patient height, weight gender and age.

The imaging protocol will be standardized for consistency of timing. Prior to the ultrasound imaging the patient and ultrasound machine will be positioned with the patient laying flat on their back with the ultrasound machine immediately next to the patient's stretcher. A numbered study identification number (ID) will be entered into the US machine instead of any actual patient identifiers. The patient will have the area of their chest and abdomen exposed where imaging will occur. No instructions will be given to the patient about the imaging other that to lay still and lay flat. The patient will not be told to take a deep breath or to hold their breath or to position themselves in any way. The study subject (i.e. physician) will stand to the left or right of the patient with the transducer in hand.

Imaging will commence when directed by research staff. The study subject (i.e. physician) is instructed to obtain a specific view of the heart as rapidly as possible, with an end goal of obtaining a clear view of the heart as it contracts. The study subject is instructed to balance speed and imaging quality, but the predominant instruction is to get it a view of the heart beating as quickly as possible. The study subject will record a 4 second digital clip of the heart and remove the transducer from the patient's skin when they are done. Upon completing the imaging of the first view the images will be scored and the subject will prepare to be timed on the second view.

The study subject (i.e. the physician) will be randomized to initially one of two views, PSL or SX. Ultrasound images will consist of a single recorded view, either subxyphoid or parasternal. The randomization will occur immediately prior to obtaining the images. Randomization will occur using binary randomization app on smart phone and this will be recorded on study sheet. The second view (whichever view was not done the first time) will be recorded immediately after the completion and recording of data from the first view.

TIMING OF CARDIAC IMAGES Timing will occur using a standardized protocol. The subject will be told to start their imaging at the direction of research staff. The timing will start when the ultrasound transducer touches the patients skin.The timing will end when the transducer is removed from the patients skin for the last time.

INTERPRETATION OF CARDIAC IMAGES Images will be rated for quality by both the subject and research staff immediately after image review. This will occur blinded to each other's rating. All ultrasound images will be recorded for later review. Ultrasound images will be rated using a 5 point imaging scale. Images will be blindly reviewed by research staff at UMASS later using the same 5 point imaging scale and categorization. Images will also be reviewed later for identification of specific cardiac landmarks including Mitral Valve, Aortic Valve, Left Ventricle and Right Ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Physicians with experience in bedside cardiac ultrasound

Exclusion Criteria:

* Unwilling to consent to study
* Appropriate ultrasound equipment not available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All physicians participating in existing ultrasound educational programs will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Timing of Ultrasound Imaging | 10 seconds
  Number of seconds from start to finish of the ultrasound imaging

SECONDARY OUTCOMES:
Quality of Ultrasound Imaging | 5 seconds
  The quality of the ultrasound images based on an ordinal numeric scale of image quality. Minimum =1 and maximum =5. Higher numbers equal better imaging quality. There is no subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD. PhD, Principal Investigator — UMASS Medical School
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be presented at scientific meetings and published in peer reviewed publications.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: available after completion of statistical review and write up of results.
Access Criteria: Freely available to whomever requests.

REFERENCES:
- [Background] Yu T, Weil MH, Tang W, Sun S, Klouche K, Povoas H, Bisera J. Adverse outcomes of interrupted precordial compression during automated defibrillation. Circulation. 2002 Jul 16;106(3):368-72. doi: 10.1161/01.cir.0000021429.22005.2e. PMID 12119255
- [Background] Steen S, Liao Q, Pierre L, Paskevicius A, Sjoberg T. The critical importance of minimal delay between chest compressions and subsequent defibrillation: a haemodynamic explanation. Resuscitation. 2003 Sep;58(3):249-58. doi: 10.1016/s0300-9572(03)00265-x. PMID 12969599
- [Background] Vaillancourt C, Everson-Stewart S, Christenson J, Andrusiek D, Powell J, Nichol G, Cheskes S, Aufderheide TP, Berg R, Stiell IG; Resuscitation Outcomes Consortium Investigators. The impact of increased chest compression fraction on return of spontaneous circulation for out-of-hospital cardiac arrest patients not in ventricular fibrillation. Resuscitation. 2011 Dec;82(12):1501-7. doi: 10.1016/j.resuscitation.2011.07.011. Epub 2011 Jul 18. PMID 21763252
- [Background] Clattenburg EJ, Wroe P, Brown S, Gardner K, Losonczy L, Singh A, Nagdev A. Point-of-care ultrasound use in patients with cardiac arrest is associated prolonged cardiopulmonary resuscitation pauses: A prospective cohort study. Resuscitation. 2018 Jan;122:65-68. doi: 10.1016/j.resuscitation.2017.11.056. Epub 2017 Nov 23. PMID 29175356
- [Background] Huis In 't Veld MA, Allison MG, Bostick DS, Fisher KR, Goloubeva OG, Witting MD, Winters ME. Ultrasound use during cardiopulmonary resuscitation is associated with delays in chest compressions. Resuscitation. 2017 Oct;119:95-98. doi: 10.1016/j.resuscitation.2017.07.021. Epub 2017 Jul 25. PMID 28754527
- [Background] Zhan L, Yang LJ, Huang Y, He Q, Liu GJ. Continuous chest compression versus interrupted chest compression for cardiopulmonary resuscitation of non-asphyxial out-of-hospital cardiac arrest. Cochrane Database Syst Rev. 2017 Mar 27;3(3):CD010134. doi: 10.1002/14651858.CD010134.pub2. PMID 28349529